CLINICAL TRIAL: NCT03412851
Title: COmparing CeNters ThRombectomy Aspiration STentretriever
Acronym: CONTRAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Alejandro González, Principal Investigator, Hospitales Universitarios Virgen del Rocío
Other Study IDs: CO-18-V1.0
Record Dates: First submitted 2018-01-12; First posted 2018-01-29 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Acute Stroke
Keywords: Thrombectomy; Stentriever; ADAPT
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A Direct Aspiration First Pass Technique
  Interventions: Other: A Direct Aspiration First Pass Technique
- Stentriever Thrombectomy
  Interventions: Other: Stentriever Thrombectomy

INTERVENTIONS:
Other: A Direct Aspiration First Pass Technique — Distal aspiration technique
  Groups: A Direct Aspiration First Pass Technique
Other: Stentriever Thrombectomy — Thrombectomy with stent retriever
  Groups: Stentriever Thrombectomy

SUMMARY:
Our aims is to evaluate the equality in efficacy and safety between direct aspiration technique and stent retriever thrombectomy procedure in anterior circulation strokes in a multicenter, prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Subject experiencing an acute ischemic stroke in which imaging demonstrates a vascular occlusion located in the distal internal carotid artery (ICA) through the distal middle cerebral artery (MCA).
* Subjects in which the aspiration technique is used for at least the first two thrombectomy passes per occluded vessel.
* Subjects older than 18 yo.
* Subjects with a prestroke modified Rankin scale of 0-2 and presenting with an NIHSS of 2-30.
* Subjects that the operator feels may be treated with endovascular therapy
* Subjects in which computed tomography (CT)/Magnetic Resonance Imaging (MRI) demonstrates an infarct size of less than 70cc on MRI or Alberta Stroke Program Early CT (ASPECTS) score overall of 6 or better.
* Subjects in which groin puncture can be obtained within 6 hours of symptom onset (with or without Total Plasminogen Activator administration). In those Patients of more than 8 hours or awake stroke or of unknown onset should be individualized the treatment and must exist area of penumbra in CT perfusion
* Subjects who have consented in accordance with local Institutional Review Board requirements

Exclusion Criteria:

* Absence of large vessel occlusion on neuroimaging.
* Platelet count < 100 x 10³ cells/mm³ or known platelet dysfunction.
* Contraindication to CT and/or MRI (i.e., due to contrast allergy or prior implant that precludes MRI imaging).
* Previously documented contrast allergy that is not amenable to medical treatment.
* Women who are pregnant or breastfeeding at time of intervention.
* Evidence of brain hemorrhage on CT and/or MRI at presenting hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke in which imaging demonstrates a vascular occlusion located in the distal internal carotid artery (ICA) through the distal middle cerebral artery (MCA).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
modified rankin scale (mRs) at 90 days [effectiveness] | 90 days
  Is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  Score Description: The scale runs from 0-6, running from perfect health without symptoms to death.
  0 No symptoms at all
  No significant disability despite symptoms; able to carry out all usual duties and activities Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance Moderate disability; requiring some help, but able to walk without assistance Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance Severe disability; bedridden, incontinent and requiring constant nursing care and attention Dead [Time Frame: 90 days]

SECONDARY OUTCOMES:
Symptomatic intracranial bleeding [safety of the technique] | First 14 days
  The rate of patients with intracranial hemorrhage (measured by computed tomography) with worsening of 4 points on the NIHSS scale will be evaluated.
Thrombolysis in cerebral infarction (TICI) scale 2b-3 [effectiveness] | Up to 24 hours after endovascular reperfusion
  After endovascular reperfusion technique, TICI score will be evaluated in all consecutive patients. The rate of TICI 2b-3 will be recorded as a effectiveness endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro González, MD, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (9):
- Spain (9):
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario, Valladolid

IPD SHARING:
Plan to Share IPD: No